CLINICAL TRIAL: NCT02057562
Title: Impact of Diverticular Disease on the Detection of Colon Adenomas
Acronym: DECADE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Peter Klare, MD, Technical University of Munich
Other Study IDs: DECADE
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Colon Adenoma; Diverticulosis
Keywords: Adenoma; Diverticular disease; Diverticulosis; Colorectal carcinoma; Polyp
MeSH Terms: conditions — Diverticulum; Adenoma; Diverticular Diseases; Colorectal Neoplasms; Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Colon polyps and mucosa
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Routine colonoscopy: Patients receiving routine colonoscopy (for a multitude of indications) at the study centers are eligible for participation

SUMMARY:
Benign adenomas of the colon have the potential to degenerate and become malignant. Therefore adenomatous polyps should be detected and resected during colonoscopy. Factors like advanced age and male gender are associated with the detection of adenomas. The same epidemiological pattern can be found with regard to colon diverticula. Furthermore, western world countries report higher incidences of both colorectal carcinoma as well as diverticular disease. It is not known whether a correlation exists between both entities. Some recent data have postulated higher adenoma detection rates in patients with concomitant diverticular disease (Rondagh EJ et al. Eur J Gastroenterol Hepatol. 2011; 23:1050-5. Kieff BJ et al. Am J Gastroenterol 2004; 99: 2007-11). If a positive correlation could be found this would possibly affect recommendations regarding colonoscopy surveillance intervals for patients with and without diverticular disease. The investigators therefore plan to conduct the following trial.

ELIGIBILITY:
Inclusion Criteria:

* indication for colonoscopy
* age >= 18 years

Exclusion Criteria:

* pregnant women
* patients denying written consent
* indication for colonoscopy: familial adenomatous polypose
* indication for colonoscopy: inflammatory bowel disease
* indication for colonoscopy: previously known colon polyp/adenoma/carcinoma
* history of colon surgery
* contraindication for resection of polyps
* American Society of Anesthesiologists (ASA) class IV, V or VI

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving routine colonoscopy at the both study centers are eligible for participation.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-02; Primary Completion 2016-09 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | up to 2 weeks (participants will be followed for the duration of hospital stay or outpatient treatment, an expected average of 2 weeks)
  After obtaining the histopathological diagnosis of resected polyps (approximately 3 days - 2 weeks after colonoscopy ) accuracy of optical diagnosis can be determined

SECONDARY OUTCOMES:
Polyp detection rate | up to one day
  a maximum of one day is expected for colonoscopy
Frequency of colon diverticulosis | up to one day
  a maximum of one day is expected for colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Peter Klare, MD, Principal Investigator — II. Medizinische Klinik, Klinikum rechts der Isar der Technischen Universität München, Germany; Peter Born, Prof. Dr., Study Chair — Innere Medizin II, Rotkreuzklinikum München, Nymphenburger Str. 163, München, Germany; Stefan von Delius, MD, Study Director — II. Medizinische Klinik, Klinikum rechts der Isar der Technischen Universität München, Germany
Locations (2):
- Germany (2):
  - Rotkreuzklinikum München, München, Deutschland
  - II Medizinische Klinik am Klinikum rechts der Isar der Technischen Universität München, München, Deutschland